CLINICAL TRIAL: NCT04458129
Title: EFFECT OF POLYETHYLENE GLYCOL TREATMENT ON INTESTINAL INFLAMMATION ASSOCIATED WITH CYSTIC FIBROSIS IN CHILDREN
Brief Title: Polyethylene Glycol and Intestinal Inflammation in Cystic Fibrosis
Acronym: MUCOLAX
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2019/25
Record Dates: First submitted 2020-06-30; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; intestinal inflammation; fecal calprotectin; microbiota; children; polyethylene glycol
MeSH Terms: conditions — Cystic Fibrosis | interventions — Therapeutics; Polyethylene Glycols

STUDY DESIGN:
Intervention Model Description: Bi-centric, non-comparative, prospective, Phase II trial according to a Fleming scheme.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Polyethylene glycol treatment (Experimental): Study participants will take a 3-month laxative treatment with polyethylene glycol for 3 months.
  Interventions: Drug: Treatment with polyethylene glycol (Macrogol 4000)

INTERVENTIONS:
Drug: Treatment with polyethylene glycol (Macrogol 4000) — 3-month treatment with polyethylene glycol (Macrogol 4000), powder for oral solution, in 4g and 10g sachets. Dosage of 0.7 g/kg/day, with a maximum dose of 20 g/day.

SUMMARY:
The main objective of the study is to evaluate the effectiveness of polyethylene glycol treatment on intestinal inflammation in children with cystic fibrosis. In this test, a method adapted from the Fleming one-step scheme will be used. The success rate is measured by the proportion of patients with fecal calprotectin levels < 250 µg/g at 3 months after treatment initiation.

DETAILED DESCRIPTION:
Cystic fibrosis is one of the most frequent serious genetic diseases in France (7000 patients). It is the consequence of mutations in the CFTR gene, encoding a protein involved in the hydro-electrolytic balance of secretions. Beyond the well-known lung damage in these patients, intestinal inflammation is present in the majority of patients.

While advances in the management of cystic fibrosis are increasing patient life expectancy, other issues are emerging, including the impact of this chronic intestinal inflammation on the nutritional status and high risk of digestive cancers (Maisonneuve, 2013; Garg and Ooi, 2017; Yamada, 2018).

Currently, no management is proposed to treat this intestinal inflammation. The use of laxatives to fluidize digestive secretions and restore a digestive ecosystem close to the healthy subject could constitute a new therapeutic approach to this intestinal inflammation, as previously shown in the mouse model of cystic fibrosis (De Lisle, 2007). However, to date, to the investigator's knowledge, no studies have evaluated the effect of laxative treatment on intestinal inflammation of cystic fibrosis in humans.

This study is a bi-centric, non-comparative, prospective study for a phase II trial according to a Fleming scheme.

Study participants will take a 3-month laxative treatment with polyethylene glycol for 3 months. In addition to the inclusion visit, a follow-up visit will take place at 3 months and 3 intermediate telephone calls will be made to ensure efficacy, tolerance and compliance.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 4 years old and <18 years old ;
* Patient with cystic fibrosis (sweat test > 60 mmol/l and/or molecular biology identifying mutations in the CFTR gene) with associated pancreatic insufficiency (fecal elastase <100 µg/g);
* With a rapid calprotectin assay result via the IBDoc test (Bühlmann®) superior or equal to 250 µg/g;
* Person affiliated or benefiting from a social security scheme;
* Free, informed and written consent signed by the holders of parental authority and the investigator before any examination required by the research and oral and/or written consent by the participant (depending on his/her age).

Exclusion Criteria:

* Ongoing processing that can modulate the functionality of the CFTR (such as lumacaftor-ivacaftor protein therapy);
* Patient already on polyethylene glycol or other laxative within 3 months before the inclusion visit;
* Patient with diarrhea at inclusion (diarrhea will be defined as the presence of 3 or more stools / day in the 7 days prior to the inclusion visit);
* Acute viral or bacterial diarrhea in the month prior to the inclusion visit (associated with fever);
* Cure of oral or intravenous antibiotics or antifungals in the month preceding the collection of samples;
* Change in background treatment in the month prior to the inclusion visit (oral or inhaled corticosteroid therapy, azithromycin, inhaled antibiotic therapy, inhaled antifungal agent, proton pump inhibitors);
* Taking probiotics in the month before the inclusion visit;
* Transplanted patient (on immunosuppressants);
* Patient with IBD or celiac disease;
* Patient with digestive perforation or risk of digestive perforation;
* Patient with ileus or suspicion of intestinal obstruction, symptomatic stenosis;
* History of hypersensitivity to macrogol or any of the excipients
* Holders of parental authority enjoying judicial protection.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Estimated)
Dates: Start 2020-07-08 (Estimated); Primary Completion 2022-04-08 (Estimated); Study Completion 2022-07-08 (Estimated)

PRIMARY OUTCOMES:
Impact of a 3-month polyethylene glycol treatment on intestinal inflammation assessed by measurement of fecal calprotectin (µg / g) by an ELISA biological test | 3 months after the inclusion visit i.e. 3 months after the initiation of treatment with polyethylene glycol
  proportion of patients with fecal calprotectin <250 µg / g measured by an ELISA test 3 months after initiation of treatment with polyethylene glycol, testifying to the absence of intestinal inflammation or slight inflammation.

SECONDARY OUTCOMES:
Evolution of the digestive inflammatory response, assessed by measurement of fecal calprotectin (µg / g) | Change from Baseline fecal calprotectin measurement at 3 months
  Evolution of the digestive inflammatory response, assessed by measurement of fecal calprotectin (µg / g) by an ELISA biological test between the initiation of treatment (D0) and 3 months of treatment with polyethylene glycol (M3)
Evolution of the digestive inflammatory response, assessed by Analysis of the expression of genes involved in the inflammatory and pro-oncogenic response | Change from Baseline measurement at 3 months
  Analysis of the expression of genes involved in the inflammatory and pro-oncogenic response, using NanoString Technology and the nCounters® PanCancer Immune Profiling Panel
Evolution of the digestive symptoms, assessed by the JenAbdomen CF-score | Change from Baseline measurement at 3 months
  The JenAbdomen CF-score has been described in the following publication Tabori H. et al. Abdominal symptoms in cystic fibrosis and their relation to genotype, history, clinical and laboratory findings. PloS One 12,e0174463 (2017).
  the JenAbdomen CF-Score is based on a CF patient-reported outcome measure (PROM) that includes all relevant gastrointestinal symptoms and their impact on subjective quality of life
Evolution of the quality of life scores, assessed by the CFQ-R questionnaire | Change from Baseline measurement at 3 months
  The CFQ-R questionnaire has been described in the following publication: Modi, A. C. & Quittner, A. L. Validation of a disease-specific measure of health-related quality of life for children with cystic fibrosis. J. Pediatr. Psychol. 28, 535-545 (2003).
  The Cystic Fibrosis Questionnaire-Revised (CFQ-R) is a disease-specific health-related quality of life (HRQOL) measure for children, adolescents and adults with cystic fibrosis (CF). It is a profile measure of HRQOL with several different domains. It has undergone extensive reliability and validity testing.
  The Cystic Fibrosis Questionnaire-Revised (CFQ-R) application calculates the score derived from the CFQ-R, on a 0-100 scale with higher scores indicating better HRQoL.
Evolution of the composition of the bacterial intestinal microbiota | Change from Baseline measurement at 3 months
  The composition of the bacterial intestinal microbiota will be assessed by High-throughput sequencing and phylogenetic allocation of the bacterial flora (on MiSeq, from Illumina®)
Evolution of the composition of the fungal intestinal microbiota | Change from Baseline measurement at 3 months
  The composition of the fungal intestinal microbiota will be assessed by high-throughput sequencing and phylogenetic allocation of the fungal flora (on MiSeq, from Illumina®)
Evolution of the pulmonary inflammation, assessed by the dosage of calprotectin in the sputum | Change from Baseline measurement at 3 months
  Evolution of the Pulmonary inflammation will be assessed by measurement of salivary calprotectin (µg / g) by an ELISA biological test between the initiation of treatment (D0) and 3 months of treatment with polyethylene glycol (M3)

CONTACTS AND LOCATIONS:
Overall Officials: Marie M MITTAINE, MD, Principal Investigator — CHU de Toulouse - Hôpital des Enfants - Centre de Ressources et de Compétences de la Mucoviscidose (CRCM) pédiatrique